CLINICAL TRIAL: NCT05533424
Title: Ultrasound Guided Quadratus Lumborum Block Versus Transversus Abdominis Plane Block as Postoperative Analgesia in Patients Undergoing Abdominal Cancer Surgery.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nevert Adel, assist. prof. of anesthesia and pain management, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: R.22.08.1787
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Abdominal Cancer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group quadratus lumborum (Active Comparator): the patient will be positioned supine with lateral tilt , and the transducer was placed at the level of the anterior superior iliac spine and moved cranially until the three abdominal wall muscles were clearly identified. The external oblique muscle was followed posterolaterally until its posterior border was visualized . The probe was tilted down to identify a bright hyperechoic line that represented the middle layer of the thoracolumbar fascia. The needle will be inserted in plane from anterolateral to posteromedial. The needle tip was placed between the thoracolumbar fascia and the QL muscle, and after negative aspiration, the correct position of the needle was proved by injection of 5 mL of normal saline to confirm the space with a hypoechoic image and hydrodissection. An injection of 20 mL of 0.25% bupivacaine was applied
  Interventions: Other: quadratus lumborum
- Group transversus abdominis plane (Active Comparator): the probe will located between the iliac crest and the lower costal margin in the anterior axillary line at the level of umbilicus, and the layers of abdominal wall were identified (external oblique, internal oblique, and transverse abdominis muscles). In-plane technique was used and the tip of the needle was inserted between the internal oblique and transverse abdominis muscles. After negative aspiration (to exclude intravascular injection), 20 mL of 0.25% bupivacaine was injected. The same technique will be performed on the other side
  Interventions: Other: transversus abdominis plane

INTERVENTIONS:
Other: quadratus lumborum — the patient will be positioned supine with lateral tilt , and the transducer was placed at the level of the anterior superior iliac spine and moved cranially until the three abdominal wall muscles were clearly identified. The external oblique muscle was followed posterolaterally until its posterior border was visualized . The probe was tilted down to identify a bright hyperechoic line that represented the middle layer of the thoracolumbar fascia. The needle will be inserted in plane from anterolateral to posteromedial. The needle tip was placed between the thoracolumbar fascia and the QL muscle, and after negative aspiration, the correct position of the needle was proved by injection of 5 mL of normal saline to confirm the space with a hypoechoic image and hydrodissection. An injection of 20 mL of 0.25% bupivacaine was applied
  Arms: Group quadratus lumborum
Other: transversus abdominis plane — the probe will located between the iliac crest and the lower costal margin in the anterior axillary line at the level of umbilicus, and the layers of abdominal wall were identified (external oblique, internal oblique, and transverse abdominis muscles). In-plane technique was used and the tip of the needle was inserted between the internal oblique and transverse abdominis muscles. After negative aspiration (to exclude intravascular injection), 20 mL of 0.25% bupivacaine was injected. The same technique will be performed on the other side
  Arms: Group transversus abdominis plane

SUMMARY:
Abdominal surgery is usually associated with severe postoperative pain. The transverse abdominal plane (TAP) block is considered an effective means for pain control in such cases. The quadratus lumborum (QL) block is another option for the management of postoperative pain.

The aim of this study is to evaluate the efficacy and safety of quadrates lumborum blocks and Transversus abdominis plane blocks for pain management after abdominal cancer surgery.

DETAILED DESCRIPTION:
Postoperative pain is severe in patients undergoing abdominal surgery, and severe pain not only affects the rate of recovery of patients but also induces a series of pathophysiological reactions. Therefore, it is very important for perioperative patients to have a safe and effective pain management model. Although classic postoperative analgesia methods can provide effective pain relief after surgery, their administration has a well-defined risk of side effects. Recently, with the rise in enhanced recovery after surgery, nerve blocks have become the key link in multimodal analgesic regimes.

As effective constituents of multimode analgesia, quadratus lumborum (QL) block and transversus abdominis plane (TAP) block are mainly used for postoperative analgesia in abdominal surgery.

Aim of this study is to compare between the analgesic effecacy of quadrates lumborum block and transverses abdominal plane block

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the study, aged 20-60 years,
* with ASA Physical Status Class I and II,
* scheduled for abdominal cancer surgery under general anesthesia

Exclusion Criteria:

* infection at injection site,
* allergy to local anesthetics,
* coagulation disorders,
* physical or mental diseases which could interfere with the evaluation of pain scores
* kidney failure or liver failure.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
The total dose of morphine | in the first 24 hours after surgery
  amount of morphine in mg

SECONDARY OUTCOMES:
visual analog score | postoperatively at 30 min and 2, 4, 6, 12, and 24 hours
  ranging from 0 to 10, where 0 no pain and 10 maximum pain
visual analog score | postoperatively 2 hours
  ranging from 0 to 10, where 0 no pain and 10 maximum pain
visual analog score | postoperatively at 4 hours
  ranging from 0 to 10, where 0 no pain and 10 maximum pain
visual analog score | postoperatively at 6 hours
  ranging from 0 to 10, where 0 no pain and 10 maximum pain
visual analog score | postoperatively at 12 hours
  ranging from 0 to 10, where 0 no pain and 10 maximum pain
visual analog score | postoperatively at 24 hours
  ranging from 0 to 10, where 0 no pain and 10 maximum pain

CONTACTS AND LOCATIONS:
Locations (1):
- Nevert Adel Abdel Ghaffar, Al Mansurah, Egypt